CLINICAL TRIAL: NCT02950090
Title: MobilWise: Mobile Phone Remote Coaching After Worksite Joint ADventure Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21AR065054-01 (NIH)
Record Dates: First submitted 2016-10-24; First posted 2016-10-31 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee symptoms; physical activity; Fitbit; Accelerometer; remote coaching
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MobilWise (Experimental): MobilWise will use data transmitted from an affordable accelerometer-based personal monitor (Fitbit Flex) via Fitabase to: allow a remote coach to view and collect physical activity data generated by the personal monitor, and use that data to formulate and provide tailored behavioral support, using motivational interviewing. The coach has a phone conversation weekly x 12 using motivational interviewing with participants to set goals and encourage activity. Coaches mention patient use of treatment elements (accountability) and will be positively reinforcing for adherent participants, or will include positive statements for those who are not adherent (supportive).Participants are also encouraged to use all the features of Fitbit (social networking, challenges, email reminders).
  Interventions: Behavioral: MobilWise
- Fitbit Only (Active Comparator): will use data transmitted from an affordable accelerometer-based personal monitor (Fitbit Flex) to monitor their own progress and physical activity level without coaching support. Participants are again encouraged to use all the features of Fitbit (social networking, challenges, email reminders) to achieve activity levels.
  Interventions: Behavioral: Fitbit Only
- Waitlist Control (No Intervention): Participants in the waitlist arm have exposure to the usual wellness supports provided by the company: Motiva is the internal corporate wellness program that is under the direction of the Chief Medical Officer. Initiated in 2000, Motiva is staffed by two full- time health professionals and two full-time healthy lifestyle professionals. Motiva provides wellness programming year round on a BCBSIL intranet web page plus an individual page called myMotiva, where self- assessment of health risks, including weight and physical activity behavior, is encouraged. Participating in myMotiva allows individuals to earn up to $200 per year in an incentive program called Wellness Rewards

INTERVENTIONS:
Behavioral: MobilWise — see arm description for MobilWise above
  Arms: MobilWise
Behavioral: Fitbit Only — see arm description for Fitbit above
  Arms: Fitbit Only

SUMMARY:
MobilWise, a worksite physical activity intervention for employees at high risk for knee osteoarthritis (OA), is being tested in a developmental randomized controlled trial at a collaborating worksite to determine if remotely- coached physical activity counseling can increase and sustain physical activity in this population. Knee osteoarthritis is a major public health problem and a leading cause of disability and work absenteeism/presenteeism in the US workforce. The overarching goal of this program is to develop and disseminate an affordable, efficient, efficacious physical activity intervention to large groups of employees at risk for knee OA. The Mobil Wise intervention is administered by health professionals, who will use data transmitted from an affordable accelerometer-based personal monitor (Fitbit Flex) via customized remote coach interface to 1) allow the remote coach to view and collect physical activity data generated by the personal monitor, and 2) use that data to formulate and provide tailored behavioral support, using motivational interviewing. This project has the potential to have a tremendous impact on improving symptoms and quality of life of persons with chronic knee pain and decreasing the functional limitation, work absenteeism/presenteeism, and soaring healthcare utilization associated with knee OA.

DETAILED DESCRIPTION:
Because the US population is aging and obesity is rising dramatically, the epidemic of arthritis-associated disability and its associated costs will significantly worsen, largely due to the consequences of knee osteoarthritis (OA). Knee OA is already a major cause of work disability and work absenteeism/presenteeism, especially among obese and overweight employees. In addition, total knee replacement surgeries have increased by 161.5% among Medicare participants over the past 20 years and are expected to quadruple in the next 20 years. Increased physical activity can relieve the pain and activity limitations of individuals with knee OA, but this healthy lifestyle behavior has not been embraced by a substantial proportion of the employed population. The overarching goal of this program is to develop and disseminate an affordable, efficient, efficacious physical activity intervention that can assist large groups of employees with or at risk for knee OA to attain and maintain healthy physical activity behavior. MobilWise is a 12-week RCT pilot that will use data transmitted from an affordable accelerometer-based personal monitor (Fitbit Flex) via customized remote- coach interface to 1) allow a remote coach to view and collect physical activity data generated by the personal monitor, and 2) use that data to formulate and provide tailored behavioral support via mobile phone, ba sed on the supportive accountability model and using motivational interviewing. The MobilWise intervention will use the media communication mode preferred by the participant (text, voice call, or video chat) to attain and sustain healthy physical activity behavior in Blue Cross Blue Shield of Illinois employees with knee symptoms after previous completion of an in-person, intensive intervention (Joint ADventure). Six month follow-up measures are planned. Specific aims are to: 1) assess the feasibility of conducting a randomized controlled trial of the Mobil Wise intervention at this worksite, 2) estimate the effectiveness of the intervention to increase objectively-measured physical activity, 3) to develop/refine the customized remote coach-interface, dashboard, and coaching protocol, and 4) to examine the accuracy of the affordable personal monitor (Fitbit Flex) by comparing that output with data from the state-of-the-art GT3X+ accelerometer. This study leverages the combined clinical and technologic expertise of Northwestern's Arthritis Center Accelerometer Unit and its Center for Behavioral Intervention Technologies, in cooperation with the Fitbit technology team and the Blue Cross Blue Shield of Illinois Corporation. If successful, a multi-site randomized controlled trial/R01 proposal will follow to demonstrate the effectiveness/cost-effectiveness of the Mobil Wise intervention in larger worksite populations. Given the influence that BCBS has in shaping future health practices and the scalability/generalizability of the proposed intervention, this research could have a tremendous impact on improving symptoms and quality of life for those with early knee OA as well as preventing the work absenteeism/presenteeism, work disability, and increased healthcare costs associated with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* 18 y/o men and women after completion of the Joint ADventure intervention (included only overweight or obese persons over age 18 with chronic knee symptoms)
* naive to Joint ADventure (no Minimum BMI) but with knee symptoms of pain, aching or stiffness on most days over the past 3 months, and have the ability to ambulate at least household distances (50ft), the ability to speak and read English.

Exclusion Criteria:

* no primary diagnosis of fibromyalgia or inflammatory arthritis
* no co-morbidity that is more functionally limiting than the knee symptoms (e.g. spinal stenosis, peripheral vascular disease or residual effects of stroke)
* no co-morbid condition (based on medical history review) that contraindicates a physical activity intervention
* no total joint re- placement surgery within the past 1 year and no plans for total joint replacement in the next 12 months
* no plans to relocate away from the Chicago-land area in the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Accelerometer counts/day; | change from baseline and 3 months
  Minutes of non-sedentary activity/day
Accelerometer counts/day; | change from baseline to 6 months
  Minutes of non-sedentary activity/day;
Accelerometer counts/day; | change from 3 months to 6 months
  Minutes of non-sedentary activity/day

SECONDARY OUTCOMES:
Fitbit measured physical activity | 6 months of study
  Minutes of non-sedentary activity/day

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided